CLINICAL TRIAL: NCT00002014
Title: A Phase I Study to Evaluate the Pharmacokinetics, Safety and Antiviral Effects of Concurrent Administration of Zidovudine (AZT) and 2'3'-Dideoxyinosine (ddI) in Patients With Human Immunodeficiency Virus (HIV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 052A; 01
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-08

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Evaluation; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To determine the safety and tolerance of various combinations of zidovudine (AZT) and didanosine (ddI) administered concurrently. To determine the pharmacokinetics of concurrent AZT and ddI administered orally. To evaluate the antiviral, immunologic and virologic effects of AZT and ddI administered concurrently.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Acyclovir not to exceed two 14-day courses of therapy during trial. Discontinue ddI while receiving acyclovir.

Patients must have the following:

* Positive HIV antibody using federally licensed ELISA test kit.
* CD4 counts < 400 on two consecutive visits within one month prior to entry.

Prior Medication:

Allowed:

* Zidovudine (AZT) if treated for less than 120 days.
* Pharmacologic doses of steroids if given for management of Pneumocystis carinii pneumonia (PCP) (not to exceed 21 days).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

- Visceral or progressive Kaposi's sarcoma (KS) (defined by > 10 new lesions in the thirty days prior to entry) or patients who require chemotherapy or radiation therapy for Kaposi's sarcoma. Other concurrent neoplasms other than basal cell carcinoma of skin or in situ carcinoma of the cervix. Malabsorption as defined by persistent diarrhea ( > 4 stools/day for four weeks) which is unresponsive to antidiarrheal agents. Opportunistic infection requiring maintenance therapy. History of Central Nervous System opportunistic infections (e.g., toxoplasmosis, cryptococcosis). History of seizure disorders. Prior history of pancreatitis. History of peripheral neuropathy or any significant signs or symptoms of neurological disease. Examinations for peripheral neuropathy should assess changes in extremities. Clinically significant hyperuricemia (tophaceous gout, urate nephropathy). History of cardiomyopathy.

Concurrent Medication:

Excluded:

* Intravenous pentamidine.
* Intravenous trimethoprim / sulfamethoxazole.
* Alcohol.
* Suppressive acyclovir therapy (see Inclusion Medications).
* Allopurinol.
* Probenecid.
* Isoniazid (INH).
* Dipyridamole.

Concurrent Treatment:

Excluded:

* Radiation therapy for Kaposi's sarcoma.

Patients with the following are excluded:

* Zidovudine (AZT) intolerance as evidenced by inability to tolerate at least 600 mg AZT daily.
* Previously intolerant to didanosine (ddI) evidenced by peripheral neuropathy or seizures or pancreatitis or gastrointestinal toxicity or hematologic toxicity.
* Diseases or conditions listed under Patient Exclusion Co-existing Conditions.

Prior Medication:

Excluded:

* Zidovudine (AZT) for > 120 days.
* Dideoxycytidine (ddC).
* Excluded within 30 days of study entry:
* Antiretroviral therapy.
* Immunomodulators.
* Biological response modifiers.
* Cytotoxic chemotherapy for Kaposi's sarcoma.
* Excluded within 60 days of study entry:
* Ribavirin.

Prior Treatment:

Excluded within 2 weeks of study entry:

* Transfusions.
* Excluded within 30 days of study entry:
* Radiation therapy for Kaposi's sarcoma.

Active substance abuse that would impair compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Univ of Miami School of Medicine, Miami, Florida
  - New England Med Ctr, Boston, Massachusetts
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Derived] Lorenzen S, Quante M, Rauscher I, Slotta-Huspenina J, Weichert W, Feith M, Friess H, Combs SE, Weber WA, Haller B, Angele M, Albertsmeier M, Blankenstein C, Kasper S, Schmid RM, Bassermann F, Schwaiger M, Liffers ST, Siveke JT. PET-directed combined modality therapy for gastroesophageal junction cancer: Results of the multicentre prospective MEMORI trial of the German Cancer Consortium (DKTK). Eur J Cancer. 2022 Nov;175:99-106. doi: 10.1016/j.ejca.2022.07.027. Epub 2022 Sep 10. PMID 36099671